CLINICAL TRIAL: NCT02249871
Title: A Trial Investigating the Influence of Omeprazole on the Pharmacokinetics of Oral Semaglutide in Healthy Subjects
Brief Title: Investigating the Influence of Omeprazole on the Pharmacokinetics of Oral Semaglutide in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-4141; 2013-005513-12 (EudraCT Number); U1111-1151-5077 (Other: WHO)
Record Dates: First submitted 2014-09-23; First posted 2014-09-26 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — semaglutide; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Semaglutide (Experimental)
  Interventions: Drug: semaglutide
- Semaglutide + Omeprazole (Experimental)
  Interventions: Drug: semaglutide; Drug: Omeprazole

INTERVENTIONS:
Drug: semaglutide — All subjects will be treated for 10 consecutive days including dose escalation, with 5 days on 5 mg oral semaglutide followed by 5 days on 10 mg oral semaglutide.
Drug: Omeprazole — Will be given daily with oral semaglutide.
  Arms: Semaglutide + Omeprazole

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the influence of omeprazole on the pharmacokinetics (the exposure of the trial drug in the body) of oral semaglutide in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18-75 years (both inclusive) at time of signing informed consent
* Body mass index of 18.5-29.9 kg/m^2 (both inclusive)
* A good general health based on medical history, physical examination, and results of vital signs, electrocardiogram and laboratory safety tests performed during the screening visit, as judged by the investigator

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using adequate contraceptive methods. Female of child bearing potential must use effective methods of birth control for the duration of the trial and for 5 weeks following last dose. Only highly effective methods of birth control are accepted (i.e., one that results in a less than 1% per year failure rate when used consistently and correctly, such as implants, injectables, combined oral contraceptives, and some intrauterine devices)
* History of Crohn's disease, ulcerative colitis, or other inflammatory bowel disease
* Hypertension (defined as sitting systolic blood pressure above or equal to 140 mmHg and/or diastolic blood pressure above or equal to 90 mmHg). If white-coat hypertension is suspected at the screening visit a repeated measurement is allowed
* Any blood draw in excess of 25 mL in the past month, or donation of blood or plasma in excess of 400 mL within the 3 months preceding screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-09-24 (Actual); Primary Completion 2015-04-01 (Actual); Study Completion 2015-04-01 (Actual)

PRIMARY OUTCOMES:
Area under the semaglutide plasma concentration time curve | From time 0 to 24 hours after the 10th daily dose

SECONDARY OUTCOMES:
Area under the SNAC plasma concentration time curve | From time 0 to 24 hours after the 10th daily dose
Number of hypoglycaemic episodes | From first dosing (Day 1) to completion of the follow-up visit (Day 43 (± 2 days))

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

REFERENCES:
- [Result] Baekdal TA, Breitschaft A, Navarria A, Hansen CW. A randomized study investigating the effect of omeprazole on the pharmacokinetics of oral semaglutide. Expert Opin Drug Metab Toxicol. 2018 Aug;14(8):869-877. doi: 10.1080/17425255.2018.1488965. Epub 2018 Jun 30. PMID 29897249
- [Derived] Overgaard RV, Navarria A, Ingwersen SH, Baekdal TA, Kildemoes RJ. Clinical Pharmacokinetics of Oral Semaglutide: Analyses of Data from Clinical Pharmacology Trials. Clin Pharmacokinet. 2021 Oct;60(10):1335-1348. doi: 10.1007/s40262-021-01025-x. Epub 2021 May 10. PMID 33969456
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com